CLINICAL TRIAL: NCT00670267
Title: An Open-Label, Dose-Escalating, Study to Evaluate the Safety, Efficacy and Tolerability of Oral Nadolol for the Treatment of Adults With Mild Asthma
Brief Title: Oral Nadolol for the Treatment of Adults With Mild Asthma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Invion, Inc. (Industry)
Collaborators: University of Houston (Other); Sandler Program for Asthma Research (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAND1002
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-04

CONDITIONS: Asthma
Keywords: Asthma; hyperresponsiveness
MeSH Terms: conditions — Asthma | interventions — Nadolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label treatment with oral Nadolol (Experimental): Dose escalation through 1.25mgs, 2.5mgs, 5.0mgs, 10mgs, 20mgs, and 40mgs of nadolol at 2 week intervals as tolerated.
  Interventions: Drug: nadolol

INTERVENTIONS:
Drug: nadolol — Nadolol, oral taken daily, doses will be escalated every two weeks over 13 weeks following a 2 week run-in.
  Other Names: Corgard

SUMMARY:
The purpose of this study is to confirm previous observations in asthmatics that chronic nadolol treatment reduces asthmatic airway hyper-responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Pre-bronchodilator FEV1 80% or greater than the predicted value.
* PC20 FEV1 ≤4 mg/ml on methacholine challenge test.
* Blood Pressure ≥ 100/65mm Hg.
* Pulse rate ≥ 60 beats/min.
* No significant health issues.
* Non-smoker or X-smoker < 10 pack/year.

Exclusion Criteria:

* History of upper/lower respiratory tract infection or asthma exacerbation within 6 weeks of first baseline visit.
* Currently diagnosed with chronic obstructive pulmonary disease (COPD).
* Used any oral or inhaled corticosteroids within 4 weeks of the first baseline visit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola A Hanania, MD, Principal Investigator — University of Houston
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Hanania NA, Singh S, El-Wali R, Flashner M, Franklin AE, Garner WJ, Dickey BF, Parra S, Ruoss S, Shardonofsky F, O'Connor BJ, Page C, Bond RA. The safety and effects of the beta-blocker, nadolol, in mild asthma: an open-label pilot study. Pulm Pharmacol Ther. 2008;21(1):134-41. doi: 10.1016/j.pupt.2007.07.002. Epub 2007 Jul 17. PMID 17703976
- [Background] Nguyen LP, Lin R, Parra S, Omoluabi O, Hanania NA, Tuvim MJ, Knoll BJ, Dickey BF, Bond RA. Beta2-adrenoceptor signaling is required for the development of an asthma phenotype in a murine model. Proc Natl Acad Sci U S A. 2009 Feb 17;106(7):2435-40. doi: 10.1073/pnas.0810902106. Epub 2009 Jan 26. PMID 19171883
- See also: ERS Publication: Response to salbutamol in patients with mild asthma treated with nadolol — http://erj.ersjournals.com/content/36/4/963.long

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label Treatment With Oral Nadolol
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Open Label: nadolol: Nadolol, oral taken daily, doses will be escalated every two weeks over 13 weeks following a 2 week run-in.
Arm/Group | Open Label
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 32.6 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Dose at Study Termination Across Participants
Description: The outcome measure describes the mean daily dose achieved by the subjects at study termination. This data includes one subject who terminated early, having reached 2.5mgs and subsequently reducing to 1.25mgs prior to dropping out.
Time Frame: Baseline to end of study (105 days)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Open Label Treatment With Oral Nadolol
Number analyzed (Participants) | 10
mg | 29.6 (16.8)

2. Primary Outcome: Daily Dose at Study Termination Across Participants
Description: The outcome measure describes the final daily dose achieved by the subjects in this study. The subjects described below who finished on less than the highest dose (i.e., 1.25, 5, and 10mgs) had all been down-titrated one dose (i.e., from 2.5, 10, and 20mgs) prior to completing the study on the dose reported.
Time Frame: Baseline to end of study (105 days)
Measure: Number; unit: participants
Arm/Group | Open Label Treatment With Oral Nadolol
Number analyzed (Participants) | 10
participants
  1.25mgs | 1
  2.5mgs | 0
  5.0mgs | 1
  10.0mgs | 1
  20mgs | 0
  40mgs | 7

3. Secondary Outcome: Change in Airway Hyper-reactivity Compared to Baseline (Change in PC20 Doubling Dose by Methacholine Challenge)
Description: Bronchoprovocation assessment was done by doubling doses of methacholine in accordance with the methodology recommended by the American Thoracic Society in the official policy statement adopted by the ATS Board of Directors, July 1999 (Guidelines for Methacholine and Exercise Challenge Testing-1999).
Time Frame: Baseline to end of study (105 days)
Population: Analysis excludes one early termination subject
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Open Label Treatment With Oral Nadolol
Number analyzed (Participants) | 9
mg/mL | 1.8 (1.3)

4. Secondary Outcome: Percent Change in FEV1% Predicted From Baseline to End of Study
Time Frame: Baseline to end of study (105 days)
Measure: Mean (Standard Deviation); unit: percent change in FEV1% predicted
Arm/Group | Open Label Treatment With Oral Nadolol
Number analyzed (Participants) | 10
percent change in FEV1% predicted | -5.9 (9.7)

5. Secondary Outcome: Change in Asthma Control Questionnaire (ACQ) Score Compared to Baseline
Description: In the E.F. Juniper Asthma Control Questionnaire, a lower number reflects better control of asthma symptoms. A positive change in ACQ score reflects a reduction in control compared to baseline; conversely, a negative change in ACQ score reflects an increase in control compared to baseline. The ACQ has 7 questions (the top scoring 5 symptoms, FEV1% pred. and daily rescue bronchodilator use). Patients are asked to recall how their asthma has been during the previous week and to respond to the symptom and bronchodilator use questions on a 7-point scale (0=no impairment, 6= maximum impairment). Clinic staff score the FEV1% predicted on a 7-point scale. The questions are equally weighted and the ACQ score is the mean of the 7 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled).
Time Frame: Baseline to end of study (105 days)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Treatment With Oral Nadolol
Number analyzed (Participants) | 10
units on a scale | 0.3 (0.7)

ADVERSE EVENTS:
Arm/Group | Open Label
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=10)
Reduced pulmonary function (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No